CLINICAL TRIAL: NCT02877615
Title: Randomized Efficacy and Safety Trial With Oral S 44819 After Recent Ischemic Cerebral Event. International, Multi-centre, Randomized, Doubleblind Placebo-controlled Phase II Study. (RESTORE BRAIN Study)
Brief Title: Efficacy and Safety Trial With S 44819 After Recent Ischemic Cerebral Event
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL2-44819-004; 2016-001005-16 (EudraCT Number); UTN number: U1111-1180-8991 (Other: WHO)
Record Dates: First submitted 2016-07-20; First posted 2016-08-24 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Post Stroke Recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- S 44819 150 mg twice a day (Experimental)
  Interventions: Drug: S 44819 150 mg twice a day
- S 44819 300 mg twice a day (Experimental)
  Interventions: Drug: S 44819 300 mg twice a day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S 44819 150 mg twice a day — One sachet of S 44819 150 mg and one sachet of placebo twice a day
  Arms: S 44819 150 mg twice a day
Drug: S 44819 300 mg twice a day — Two sachets of S 44819 150 mg twice a day
  Arms: S 44819 300 mg twice a day
Drug: Placebo — Two sachets of placebo twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of S 44819 in enhancing functional recovery after an ischemic stroke.

ELIGIBILITY:
Inclusion criteria :

* Patients aged between 18 and 85 years (both inclusive)
* Acute ischemic stroke that occured between 72 hours (3 days) and 192 hours (8 days) (both inclusive) before inclusion

Exclusion criteria :

* Any non-selection criteria, which could have occurred after the selection visit
* Positive urinary or blood pregnancy test (for female patients of child bearing potential)
* Any clinically significant findings from the local laboratory test likely to interfere with the ability to participate in the study and / or with the study outcome
* Severe renal impairment detected in the local laboratory test
* Severe hepatic impairment or liver enzymes abnormalities found in the local laboratory test
* Stroke due to cerebral venous thrombosis
* Brain MRI showing a severe microangiopathy
* Brain imaging showing an acute haemorrhagic stroke or a symptomatic haemorrhagic transformation of the brain infarct
* Qualifying ischemic cerebral event older than 192 hours at inclusion
* Any clinically relevant abnormalities detected during the examinations likely to interfere with study procedures or study outcome,
* Repeated prolongation of ECG QTcF
* Patient or authorised representative refusing to attend study visits or to take part in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | Up to 90 days

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) total score | Selection visit Day 0 Day 5 Day 30 Day 60 Day 90 Day 105
  Efficacy criterion
Barthel Index (BI) total score | Day 30 Day 60 Day 90 Day 105
  Efficacy criterion
Montreal Cognitive Assessment scale (Moca) total score | Day 30 Day 90
  Efficacy criterion
Trail Making Test (TMT) time for part A | Day 30 Day 90
  Efficacy criterion
Adverse events | Through study completion, an average of 3 months
  Safety criterion
Suicidal ideation and suicidal behavior using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Day 5 Day 30 Day 60 Day 90 Day 105
  Safety criterion
Body weight | Selection visit Day 30 Day 60 Day 90 Day 105
  Safety criterion
Vital signs (supine for Systolic and Diastolic Blood Pressure) | Selection visit Day 0 Day 5 Day 30 Day 60 Day 90 Day 105
  Safety criterion
12 lead-ECG | Day 0 Day 5 Day 30 Day 60 Day 90 Day 105
  Safety criterion
Trail Making Test (TMT) time for part B | Day 30 Day 90
  Efficacy criterion

CONTACTS AND LOCATIONS:
Locations (121):
- Australia (10):
  - Royal Adelaide Hospital Department of Neurology, Adelaide
  - Sunshine Coast Hospital, Birtinya
  - Monash Medical Centre Department of Neurology, Clayton
  - Lyell McEwin Hospital Neurology Department, Elizabeth Vale
  - Gosford Hospital Neurosciences Department, Gosford
  - Austin Health Neurology Department, Heidelberg
  - Royal Brisbane & Women's Hospital Department of Neurology, Herston
  - Alfred Health, Melbourne
  - Royal Melbourne Hospital Department of Neurology, Parkville
  - Gold Coast University Hospital, Southport
- Belgium (7):
  - AZ Sint-Lucas Neurologie, Bruges
  - AZ. St. Jan, Bruges
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Jessa Ziekenhuis Dienst Neurologie, Hasselt
  - UZ Leuven Campus Gasthuisberg, Leuven
  - Les Cliniques Saint-Joseph, Liège
  - Sint Andries Ziekenhuis Dienst Neurologie, Tielt
- Brazil (10):
  - Hospital das Clinicas da Faculdade de Medicina de Botucatu, Botucatu
  - Clínica Neurológica e Neurocirúrgica de Joinville, Joinville
  - Hospital Carlos Fernando Malzone Departamento de Neurologia, Matão
  - IMV Pesquisa Neurológica Setor de Pesquisa Clinica, Porto Alegre
  - Hospital Sao Lucas da Pontificia Universidade Catolica RS Setor de Pesquisa Clínica, Porto Alegre
  - Hospital das Clinicas da Fac. de Med. de Ribeirao Preto Unidade de Emergencia - Centro de Estudo, Ribeirão Preto
  - Hospital das Clinicas da Fac. de med. de Ribeirao Preto Unidade de Emergiancia, Ribeirão Preto
  - Hospital Quinta D'or Departamento de Neurologia, Rio de Janeiro
  - Irmandade Santa Casa de Misericordia de Sao Paulo Ambulatório de Neurologia, São Paulo
  - UNIFESP - Universidade Federal de Sao Paulo Centro de Pesquisa em Neurologia, São Paulo
- Canada (4):
  - University of Alberta, Edmonton
  - Charles LeMoyne Hospital-CISSS de la Monteregie-Centre, Greenfield Park
  - Montreal General Hospital, Montreal
  - Saint John Regional Hospital, Saint John
- Czechia (4):
  - Fakultni nemocnice Brno Neurologicka klinika, Brno
  - Fakultni nemocnice u sv. Anny Neurologicka klinika, Brno
  - Nemocnice Jihlava, Jihlava
  - Vseobecna fakultni nemocnice II. interni klinika VFN a 1. LF UK, Prague
- France (9):
  - CHU Bdx-Hôpital Pellegrin-Tripode Service de Neurologie, Bordeaux
  - Hôpital Sud-Francilien Unité Neurovasculaire, Corbeil-Essonnes
  - CHU Henri Mondor Service de Neurologie, Créteil
  - CHU de Bicêtre Service de neurologie, Le Kremlin-Bicêtre
  - CHRU-Hôpital Roger Salengro Service de Neurologie, Lille
  - CHU-Hôpital Gui de Chaulliac Unité de Neuropshysiologie Clinique, Montpellier
  - Hôpital Lariboisière, Fernand-Vidal Service de Neurologie, Paris
  - Hôpital Sainte-Anne Service de Neurologie, Paris
  - CHU-Hôpital de la Milétrie Service de Neurologie, Poitiers
- Germany (10):
  - Klinikum Altenburger Land GmbH Neurologische Klinik, Altenburg
  - Neurologische Klinik GmbH, Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Klinikum Neukölln Klinik für Neurologie mit Stroke Unit, Berlin
  - Universitätsklinikum Erlangen Neurologische Klinik, Erlangen
  - Universitaetsklinikum Essen Neurologische Universitätsklinik Essen, Essen
  - Universitätsmedizin der Johannes Gutenberg-Universität Klinik und Poliklinik für, Mainz
  - Johannes Wesling Klinik Minden Klinik für Neurologie, Minden
  - Kreisklinikum Siegen Klinik fuer Neurologie, Siegen
  - Universitätsklinik der Eberhard-Karls Universtiät Tübingen Hertie-Institut für Klinische Hirnforschung, Tübingen
  - Universitätsklinikum Ulm Neurologische Klinik (RKU), Ulm
- Hungary (14):
  - Semmelweis Egyetem Neurologiai Klinika, Budapest
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet Neurologiai Osztaly, Budapest
  - Szent Janos Korhaz Neurologiai osztaly, Budapest
  - Honved Korhaz Stroke reszleg, Budapest
  - Orszagos Idegsebeszeti Tudomanyos Intezet, Budapest
  - Petz Aladar Megyei Oktato Korhaz Neurologiai Osztaly, Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz Neurologiai Osztaly, Kaposvár
  - Flor Ferenc Korhaz Neurologia, Kistarcsa
  - B-A-Z Megyei Korhaz es Egyetemi Oktato Korhaz Stroke, Er- es Neurologiai, Toxikologiai Osztaly, Miskolc
  - Kanizsai Dorottya Korhaz Neurologiai Osztaly, Nagykanizsa
  - Josa Andras Oktatokorhaz Neurologiai Osztaly, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont Neurologiai Klinika, Pécs
  - Soproni Erzsebet Oktato Korhaz Neurologiai Osztaly, Sopron
  - Szegedi Tudomanyegyetem Szent-Gyorgy Albert Klinikai Kozpont, Szeged
- Italy (6):
  - Vito FAZZI U.O. semplice Stroke Unit, Lecce
  - Ospedale San Giuseppe UOC di Neurologia e Stroke Unit, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale Sacro Cuore Don Calabria Negrar NEUROLOGY DEPT, Negrar
  - Istituto Neurologico mediterraneo NEUROMED Dipartimento di Medicina Riabilitativa e Specialistica Repar, Pozzilli
  - Policlinico Umberto I Emergency Department Stroke Unit, Rome
- Netherlands (5):
  - Zuyderland Medisch Centrum Afdeling Neurologie, Heerlen
  - UMC St Radboud Afdeling Neurologie, Nijmegen
  - Canisius Wilhelmina Ziekenhuis Afdeling Neurologie, Nijmegen
  - Erasmus MC Afdeling Neurologie, Rotterdam
  - Isala Klinieken Afdeling Neurologie, Zwolle
- Poland (9):
  - Samodzielny Publiczny Wojewodzki Szpital Specjalistyczny Oddzial Neurologiczny i Oddzial Udarowy, Chełm
  - M. Kopernika Provincial Specialist Hospital Dpt of Neurology, Gdansk
  - Szpital Specjalistyczny sw. Lukasza Oddzial Neurologii i Oddzial Udarowy, Gmina Końskie
  - Samodzielny Publiczny Szpital Kliniczny nr7 SUM w Katowicach Oddzial Neurologii z Pododdzialem Udarowym, Katowice
  - Miejskie Centrum Medyczne Jonscher Szpital Dr K. Jonschera, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie Oddzial Neurologii, Lublin
  - Wojewodzki Szpital Specjalistyczny SPZOZ nr 3 w Rybniku, Rybnik
  - Szpital Specjalistyczny Ducha Swietego w Sandomierzu Oddzial Neurologii, Sandomierz
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
- South Korea (7):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Medical Center Department of Neurology, Busan
  - Kyungpook National University Hospital Department of Neurology, Daegu
  - Chonnam National University Hospital Department of Neurology, Gwangju
  - Seoul National University Bundang Hospital Department of Orthopaedic, Seongnam
  - Kyung Hee University Hospital, Seoul
  - ASAN Medical Center Department of Neurology, Seoul
- Spain (12):
  - H. General de Albacete Servicio de Neurología, Albacete
  - H. Germans Trias I Pujol Servicio de Neurología, Badalona
  - H. del Mar Neurología, Barcelona
  - H. Valle de Hebrón Servicio de Neurología, Barcelona
  - H. Clinic de Barcelona Comprehensive Stroke Center, Barcelona
  - Hospital Universitari de Bellvitge Servicio de Neurología-Unidad de Ictus-Planta 9, Barcelona
  - H. Universitario de Donosti Servicio de Neurología, Donostia / San Sebastian
  - H. Josep Trueta Servicio de Neurología, Girona
  - H. Universitario La Princesa Servicio de Neurología, Madrid
  - H. Ramón y Cajal Servicio de Neurología, Madrid
  - H. Virgen del Rocío Servicio de Neurología, Seville
  - Hospital Universitario La Fe Servicio de Neurología, Valencia
- Sweden (5):
  - Hassleholms Sjukhus Stroke- och rehabiliteringsavdelningen 9, Hässleholm
  - University Hospital Department of Neurology, Linköping
  - Skaraborgs Sjukhus Skovde Strokenheten, Skövde
  - Danderyds Sjukhus Medicinmottagningen, Stockholm
  - Akademiska Sjukhuset Strokeavdelningen 85B, Uppsala
- United Kingdom (9):
  - Royal United Hospital Older People's Unit, Bath
  - Queen Elizabeth University Hospital, Glasgow
  - Northwick Park Hospital Neurology, Harrow
  - Leicester Royal Infirmary Dpt of Neurology, Leicester
  - St George's University Hospitals Stroke Research office, London
  - Nottingham City Hospital, Nottingham
  - Poole NHS Foundation Trust Stroke Unit, Poole
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield
  - Royal Stoke University Hospital Stroke Team Office, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com

REFERENCES:
- [Background] Chabriat H, Bassetti CL, Marx U, Picarel-Blanchot F, Sors A, Gruget C, Saba B, Wattez M, Audoli ML, Hermann DM. Randomized Efficacy and Safety Trial with Oral S 44819 after Recent ischemic cerebral Event (RESTORE BRAIN study): a placebo controlled phase II study. Trials. 2020 Feb 3;21(1):136. doi: 10.1186/s13063-020-4072-2. PMID 32014032
- [Result] Chabriat H, Bassetti CL, Marx U, Audoli-Inthavong ML, Sors A, Lambert E, Wattez M, Hermann DM; RESTORE BRAIN study investigators. Safety and efficacy of GABAA alpha5 antagonist S44819 in patients with ischaemic stroke: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2020 Mar;19(3):226-233. doi: 10.1016/S1474-4422(20)30004-1. PMID 32085836
- See also: Scientific publication — https://www.ncbi.nlm.nih.gov/pubmed/32085836
- See also: Scientific publication — https://www.ncbi.nlm.nih.gov/pubmed/32014032
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/